CLINICAL TRIAL: NCT01080976
Title: Comparing Google With A Focused Diabetes Search Engine
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Charles Safran, Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2009P000356
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Primary Care Physicians
- Diabetologists

SUMMARY:
Abstract Diabetes behavior can be influenced by patients exploring diabetes topics that may lack scientific credibility. The question this study examines is whether a Google or Health on the Net (HON) internet search, presents websites that would incline a more or less likely recommendation to patients ? A preliminary trial suggests that referrers recommend websites based on rules that may prioritize website source over content. This study will qualitatively assess the rules that participants use in deciding which websites are more suitable than others.

Method The investigators will inject a diabetes related search term into a HON and a Google search engine. The top 5 mutually exclusive websites from each search engine will be presented to 5 people from three groups stratified across endocrinologists, informaticians and PCPs. Participants will rank the websites and then identify the rules that they applied to reach their decision.

ELIGIBILITY:
Inclusion Criteria:

* physician, informatician, diabetologist

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Physicians, Informaticians, Diabetologists
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Safran, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Charles Safran, Brookline, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care Physicians | Diabetologists
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care Physicians | Diabetologists | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Website Ranking
Description: Primary care and diabetes clinicians' preference in a set of webpage search results on a visual analog scale (1-100) with 1 being the lowest preference and 100 being the highest. Rankings based on qualitative measures, such as perceived clinical relevance, perceived accuracy of content, and perceived timeliness of content.
Time Frame: Immediate
Population: Participants were asked to rank 10 pages of website search results from Google and HoN search engines based on clinician preference. Clinicians were further asked for feedback and opinions on how they determined their ranking. Rankings of individual websites were done by visual analog scale, from 1-100, with 100 indicated as highly preferred.
Measure: Number; unit: units on a scale
Groups:
- Primary Care Physicians: Doctors from General Practice
- Diabetologists: Doctors Specialized in Diabetes
Arm/Group | Primary Care Physicians | Diabetologists
Number analyzed (Participants) | 5 | 5
units on a scale | NA — Data no longer available due to PI (Reti S) leaving BIDMC after completion of his fellowship. PI is no longer in the United States and cannot be reached. | NA — Data no longer available due to PI (Reti S) leaving BIDMC after completion of his fellowship. PI is no longer in the United States and cannot be reached.

2. Primary Outcome: Search Engine Preference
Description: Based on the results of primary outcome 1 (Website Ranking), preference for search engine was measured qualitatively between Google and Health-on-the-Net.
Time Frame: Immediate
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care Physicians | Diabetologists
Number analyzed (Participants) | 5 | 5
Participants | NA — No data available. No record exists of this data being collected. PI (Reti S) no longer employed by BIDMC having finished the fellowship program. | NA — No data available. No record exists of this data being collected. PI (Reti S) no longer employed by BIDMC having finished the fellowship program.

ADVERSE EVENTS:
Arm/Group | Primary Care Physicians | Diabetologists
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No